CLINICAL TRIAL: NCT02703077
Title: Endoscopic Treatment of Difficult Bile Duct Stones: Use of Direct Visualization System ("Spyglass Direct Visualization System") Associated With Electrohydraulic Lithotripsy (EHL) X Hydrostatic Balloon Dilation of the Major Duodenal Papilla
Brief Title: Endoscopic Treatment of Difficult Bile Duct Stones: Spyglass + EHL x Balloon Dilation of the Papilla
Acronym: EHL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0784/10
Record Dates: First submitted 2016-02-29; First posted 2016-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-02

CONDITIONS: Common Bile Duct Gallstones; Choledocholithiasis
MeSH Terms: conditions — Gallstones; Choledocholithiasis | interventions — Sphincterotomy, Transduodenal; Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: ERCP + Spyglass + EHL (Active Comparator): This group after the diagnosis of difficult bile duct stones, will be submitted to spyglass cholangioscopy + EHL (electrohydraulic lithotripsy)
  Interventions: Procedure: Spyglass; Procedure: EHL (electrohydraulic lithotripsy); Procedure: ERCP (Endoscopic retrograde cholangiopancreatography)
- 2: ERCP + Balloon Dilation (Active Comparator): This group after the diagnosis of difficult bile duct stones, will be submitted to Balloon dilation of the papilla
  Interventions: Procedure: Balloon dilation of the papilla; Procedure: ERCP (Endoscopic retrograde cholangiopancreatography)

INTERVENTIONS:
Procedure: Spyglass — Endoscopic direct view of the bile ducts
  Other Names: Cholangioscopy; Direct view cholangioscopy
  Arms: 1: ERCP + Spyglass + EHL
Procedure: Balloon dilation of the papilla — Using a hidrostatic balloon the major papilla will be dilated to facilitate the stone removal
  Other Names: Sphincteroplasty
  Arms: 2: ERCP + Balloon Dilation
Procedure: EHL (electrohydraulic lithotripsy) — With a probe a direct view lithotripsy will be performed
  Arms: 1: ERCP + Spyglass + EHL
Procedure: ERCP (Endoscopic retrograde cholangiopancreatography) — Endoscopic procedure to identify and treat biliary diseases

SUMMARY:
This study compare 2 techniques to treat difficult bile duct stones endoscopically

DETAILED DESCRIPTION:
Before enrollment of the patients into the study, the two investigators, EGHM and TAPF, will perform 10 complete cases each of ERCP (Endoscopic retrograde cholangiopancreatography) + SPYGLASS + EHL, to get more experience with the methods.

This will be a comparative study of methods, prospective, randomized study assessing the successful removal of bile duct stones considered to be difficult between the two proposed methods. A total of 100 patients will be recruited, according to the criteria for inclusion / exclusion of Appendix I. Randomization will be performed using a computer generated system. Fifty patients will be distributed in group 1 (Spyglass + electrohydraulic lithotripsy) and fifty in group 2 (with hydrostatic balloon dilation of the papilla with a extractor balloon sweep). Endoscopic retrograde cholangiopancreatography (ERCP) will be performed, and after the diagnosis of difficult stone, will be followed by randomization between the two proposed methods. In group 1, the examination with the Direct Visualization System of Bile Ducts ("Spyglass Direct Visualization System") will be held soon after the diagnosis of difficult stone and partial endoscopic papillotomy. After access to the biliary duct with the system described, and the visualization of the stone, it will be introduced gently through the working channel of a spyglass the probe to perform the electrohydraulic lithotripsy. When the fragmentation is complete the system spyglass will be removed and the pieces of stone are removed by conventional endoscopic methods. In group 2, after the diagnosis of difficult calculi and performing the partial endoscopic papillotomy, the papilla (as with papillotomy) will be dilated with a hydrostatic balloon until the maximum size allowed by the diameter of common bile duct, followed by scanning with extractor balloon. In both groups, the stone clearance will be confirmed using Spyglass cholangioscopic exploration of the bile duct. In case of failure in stone removal by some of the methods studied, it will be performed biliary drainage with plastic stent.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Able to give consent
* Submitted to the examination of endoscopic retrograde cholangiopancreatography (ERCP), with identification of stones in the bile duct considered difficult.
* Agreed and signed the Term of Consent.

Exclusion Criteria:

* Age below 18 years
* Incapable of giving consent
* Pregnant
* Gastrointestinal bypass surgery with previous reconstructions as a Billroth II or Roux-en-Y
* Patients with signs of severe acute cholangitis requiring biliary drainage with fast plastic stent and minimal or no contrast infusion
* Patients with previous liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-12 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Success of the intervention | intraoperative
  Defined as complete stone removal of the bile duct

SECONDARY OUTCOMES:
Time | intraoperative
  From ERCP diagnosis to end of procedure (in minutes)
Adverse events | One week
  All procedure related adverse events
X-ray time | intraoperative
  From ERCP diagnosis to end of procedure in minutes
Difficulties | intraoperative
  Procedure related technique difficulties (operator subjective evaluation) : papilla dilation, Spyglass insertion into bile duct, lithotripsy probe introduction, EHL

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Moura, PhD, Study Director — University of Sao Paulo Medical School
Locations (1):
- Endoscopy Unit - Clinics Hospital University of Sao Paulo Medical School, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Decision during trial

REFERENCES:
- [Background] Moura EG, Franzini T, Moura RN, Carneiro FO, Artifon EL, Sakai P. Cholangioscopy in bile duct disease: a case series. Arq Gastroenterol. 2014 Jul-Sep;51(3):250-4. doi: 10.1590/s0004-28032014000300015. PMID 25296087
- [Background] Attam R, Freeman ML. Endoscopic papillary large balloon dilation for large common bile duct stones. J Hepatobiliary Pancreat Surg. 2009;16(5):618-23. doi: 10.1007/s00534-009-0134-2. Epub 2009 Jun 24. PMID 19551331
- [Background] Stefanidis G, Christodoulou C, Manolakopoulos S, Chuttani R. Endoscopic extraction of large common bile duct stones: A review article. World J Gastrointest Endosc. 2012 May 16;4(5):167-79. doi: 10.4253/wjge.v4.i5.167. PMID 22624068
- [Background] Trikudanathan G, Navaneethan U, Parsi MA. Endoscopic management of difficult common bile duct stones. World J Gastroenterol. 2013 Jan 14;19(2):165-73. doi: 10.3748/wjg.v19.i2.165. PMID 23345939
- [Background] Trikudanathan G, Arain MA, Attam R, Freeman ML. Advances in the endoscopic management of common bile duct stones. Nat Rev Gastroenterol Hepatol. 2014 Sep;11(9):535-44. doi: 10.1038/nrgastro.2014.76. Epub 2014 May 27. PMID 24860928